CLINICAL TRIAL: NCT06719687
Title: Self-driving Robotic-assisted Bronchoscopy for the Diagnosis of Peripheral Pulmonary Lesions
Brief Title: Sd-RAB for the Diagnosis of PPLs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KS24054
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Pulmonary Lesions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with peripheral pulmonary lesions (Experimental): 30 patients with peripheral pulmonary lesions who meet the inclusion and exclusion criteria will be prospectively enrolled. Self-driving robotic-assisted bronchoscopy will be performed to diagnose the lesions.
  Interventions: Device: Self-driving robotic-assisted bronchoscope

INTERVENTIONS:
Device: Self-driving robotic-assisted bronchoscope — All procedures will be performed under general anesthesia with endotracheal intubation and mechanical ventilation. The self-driving robotic-assisted bronchoscope will automatically advance through airway to the target lesion according to the preoperative planning path under the guidance of electromagnetic navigation. After that, the bronchoscopist will use radial endobronchial ultrasound (rEBUS) to confirm the lesion localization. The choice of biopsy tools (eg. forceps, needles, brush, etc.) will be left to the discretion of the bronchoscopist.

SUMMARY:
This is a single-center, prospective, and single-arm study. The purpose of this study is to evaluate the feasibility and safety of a new self-driving robotic-assisted bronchoscopic system for the diagnosis of peripheral pulmonary lesions.

DETAILED DESCRIPTION:
Self-driving robotic-assisted bronchoscope (Shanghai MicroPort MedBot (Group) Corporation Limited, China) is a new robotic-assisted bronchoscopic system that can automatically advance through airway according to the preoperative planning path under the guidance of electromagnetic navigation. It can also be controlled manually by the operator. In this study, 30 patients will be prospectively enrolled to evaluate the feasibility and safety of this new self-driving robotic-assisted bronchoscopic system for the diagnosis of peripheral pulmonary lesions. The primary endpoint of this study is the complication rate. The secondary endpoints include navigation success rate, diagnostic yield, rate of rEBUS confirmation, total examination time, navigation time, and duration of finding lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years old.
2. Chest imaging shows the presence of peripheral pulmonary lesions (defined as those lesions that are surrounded by pulmonary parenchyma and located below the segmental bronchus), which are suspected to be malignant and require a non-surgical biopsy.
3. Patients have good medical adherence and signed informed consent.

Exclusion Criteria:

1. Contraindications for bronchoscopy.
2. Presence of concomitant endobronchial lesion during the bronchoscopy procedure.
3. The investigators believe that patient has other conditions that are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Complication rate | 1 month
  The complications refer to the total of device or procedure related adverse events during or within 1 month after the operation.

SECONDARY OUTCOMES:
Navigation success rate | 1 month
  Navigation success is defined as confirmation of the target lesion under rEBUS or a bronchoscope tip-to-virtual lesion distance <2 cm that allows lesion sampling. Cases in which a malignant or specific benign diagnosis is obtained are also considered as navigation success.
Diagnostic yield | 1 month
  Diagnostic yield of self-driving robotic-assisted bronchoscopy for peripheral pulmonary lesions.
Rate of rEBUS confirmation | During the procedure
  rEBUS confirmation is defined as visualization of target lesion using rEBUS during the procedure.
Total examination time | During the procedure
  Total examination time is defined from the time that the bronchoscope is inserted beyond the glottis, until the bronchoscope has been removed from the glottis after examination.
Navigation time | During the procedure
  Navigation time is defined as the time from the start of the self-driving robotic-assisted bronchoscope advancing under the guidance of electromagnetic navigation to the insertion of the ultrasound probe.
Duration of finding lesions | During the procedure
  Duration of finding lesions is defined from the insertion of the ultrasound probe to the withdrawal of the ultrasound probe.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China